CLINICAL TRIAL: NCT03834883
Title: Novel Approaches for Minimizing Drug-Induced QT Interval Lengthening: Reducing the Risk of Drug-Induced QT Interval Lengthening in Women
Brief Title: Reducing the Risk of Drug-Induced QT Interval Lengthening in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other); Purdue University (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Professor, College of Pharmacy, Purdue University, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1806935117
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Long QT Syndrome; Abnormalities, Drug-Induced
MeSH Terms: conditions — Long QT Syndrome; Abnormalities, Drug-Induced | interventions — Progesterone; ibutilide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Postmenopausal women: Progesterone (Experimental): Subjects will receive treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Interventions: Drug: Progesterone; Drug: Ibutilide
- Postmenopausal women: Placebo (Placebo Comparator): Subjects will receive oral placebo, two capsules once daily every evening for 7 days
  Interventions: Drug: Ibutilide
- Premenopausal women: Progesterone (Experimental): Subjects will receive treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Interventions: Drug: Progesterone; Drug: Ibutilide
- Premenopausal women: Placebo (Placebo Comparator): Subjects will receive oral placebo, two capsules once daily every evening for 7 days
  Interventions: Drug: Ibutilide

INTERVENTIONS:
Drug: Progesterone — Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Arms: Postmenopausal women: Progesterone; Premenopausal women: Progesterone
Drug: Ibutilide — Ibutilide 0.003 mg/kg administered to all subjects to moderately lengthen the QT interval
  Other Names: Corvert

SUMMARY:
This research will determine if oral progesterone attenuates drug-induced QT interval lengthening in a) Postmenopausal women 50 years of age or older, and b) Premenopausal women studied during the ovulation phase of the menstrual cycle. This investigation will consist of two concurrent prospective, randomized, double-blind, placebo-controlled crossover-design studies in a) Postmenopausal women, and b) Premenopausal women. Each subject will take progesterone or placebo capsules for 1 week. After a two-week "washout" (no progesterone or placebo) each subject will then take the alternative therapy (progesterone or placebo) for 1 week. After 7 days of each treatment, subjects will present to the clinical research center to receive a small dose of the QT interval-lengthening drug ibutilide, and the effect on the QT, J-Tpeak and Tpeak-Tend intervals during the progesterone and placebo phases will be compared

DETAILED DESCRIPTION:
Torsades de pointes (TdP) is a catastrophic arrhythmia associated with corrected QT (QTc) interval prolongation, which can be induced by > 150 commonly prescribed drugs. TdP risk is higher in women and is modulated by the ratio of serum progesterone and estradiol; the higher the serum progesterone and progesterone:estradiol ratio, the lower the risk, and vice-versa. TdP risk increases with age, likely due to declining postmenopausal progesterone concentrations. Methods to reduce TdP risk in postmenopausal women requiring therapy with QTc interval-prolonging drugs have not been developed. In addition, the differential effects of progesterone on drug-induced lengthening of early vs late ventricular repolarization in humans are unknown. The investigators have previously shown that oral progesterone attenuates QTc interval lengthening in young women during the menses phase when serum estradiol concentrations are low. However, whether oral progesterone remains effective for attenuating drug-induced QTc interval lengthening during menstrual cycle phases with higher serum estradiol concentrations is unknown. The efficacy of oral progesterone for attenuating drug-induced QTc interval lengthening in postmenopausal women is also unknown. Specific Aim1: Determine the efficacy of oral progesterone as a preventive method to diminish drug-induced QTc interval lengthening in postmenopausal women. Specific Aim 2: Determine the influence of oral progesterone on drug-induced lengthening of early versus late ventricular repolarization in postmenopausal women. Specific Aim 3: Determine the efficacy of oral progesterone to diminish drug-induced QTc interval lengthening in premenopausal women during the ovulation phase of the menstrual cycle, when serum estradiol concentrations are high. Specific Aim 4: Specific Aim 4: Determine the influence of oral progesterone on drug-induced lengthening of early versus late ventricular repolarization in premenopausal women during the ovulation phase of the menstrual cycle, when serum estradiol concentrations are high.

Concurrent prospective, randomized, double-blind, placebo-controlled two-way crossover-design studies will be conducted in a) Postmenopausal women > 50 years of age (n=20) and b) Premenopausal women 21-40 years of age (n=20) who will be studied during the ovulation phase of the menstural cycle. QTc interval response to low-dose ibutilide will be assessed. Subjects will receive, in randomized order (with a minimum two-week washout phase) oral progesterone 400 mg or placebo once daily for 7 days. On the morning after the 7th dose, subjects will present to the Indiana Clinical Research Center to receive one dose of the QT interval-lengthening drug ibutilide 0.003 mg/kg, after which ECGs and blood for determination of serum ibutilide concentrations will be obtained serially for 8 hours. Primary outcome measures: 1) Baseline (pre-ibutilide) Fridericia (QTFrid) and Framingham (QTFram)-corrected QT intervals, 2) Maximum QTFrid and QTFram intervals following ibutilide, 3) Maximum % change in QTFrid and QTFram intervals following ibutilide, 4) Area under the QTFrid and QTFram interval-time curves from 0-1 and 0-8 hours. Secondary outcome measures: 1) J-Tpeak interval, 2) Tpeak-Tend interval, and 5) Incidence of progesterone and ibutilide adverse effects. These studies will establish oral progesterone as a safe and effective method of attenuating drug-induced QTc interval lengthening in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women:

* 50 years of age or older
* No menstrual periods for 365 days or longer

Premenopausal women:

- 21-40 years of age

Exclusion Criteria:

* History of breast, uterine or ovarian cancer
* History of hysterectomy and/or ovariectomy
* Weight > 135 kg
* Serum K+ < 3.6 mEq/L;
* Serum Mg2+ < 1.8 mg/dL;
* Hematocrit < 26%;
* Hepatic transaminases > 3x upper limit of normal;
* Baseline Bazett's-corrected QT interval > 450 ms
* Taking hormone replacement therapy
* Diagnosis of heart failure
* Symptoms associated with heart failure:

  * Pitting edema > 2+
  * Crackles or rales on lung auscultation
  * S3 or S4 heart sounds
  * Unable to climb at least 2 flights of stairs without becoming short of breath
* Current ECG rhythm of atrial fibrillation or other tachyarrhythmia
* Family or personal history of long-QT syndrome or sudden cardiac death not associated with acute myocardial infarction
* Concomitant use of any QTc interval-prolonging drug.
* Permanently paced ventricular rhythm
* Pregnancy
* Using any hormonal contraceptives [oral contraceptives, hormone-secreting intrauterine devices (IUDs), hormonal implants]

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal - 50 years of age or older and no menstrual period for 365 days or longer
  Premenopausal - 21-40 years of age
Enrollment: 27 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Purdue University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a) Indiana CTSI ALL IN for Health Research database, and b) advertisements on the Indiana University-Indianapolis and Purdue University campuses
Pre-assignment Details: Premenopausal women: n=222 participants assessed for eligibility; n=20 consented, n=202 excluded (n=50 did not meet inclusion criteria, n=152); n=18 enrolled
  Postmenopausal women: Target sample size n=16. Did not achieve target because of delays/problems due to COVID-19 and limited budget. n=22 were assessed for eligibility; n=12 consented; 3 excluded because QTc > 450 ms; 9 enrolled; 2 dropped out in pandemic, completed 1 phase
Groups:
- Premenopausal Women: Progesterone Then Placebo; Postmenopausal Women: Progesterone Then Placebo: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days. After a two-week washout period, participants received oral placebo, two capsules once daily every evening for 7 days.
- Premenopausal Women: Placebo Then Progesterone; Postmenopausal Women: Placebo Then Progesterone: Participants received oral placebo, two capsules once daily every evening for 7 days. After a two-week washout period, participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days.
Period: First Treatment
Arm/Group | Premenopausal Women: Progesterone Then Placebo | Premenopausal Women: Placebo Then Progesterone | Postmenopausal Women: Progesterone Then Placebo | Postmenopausal Women: Placebo Then Progesterone
Started | 9 | 9 | 3 | 6
Completed | 9 | 9 | 3 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Treatment
Arm/Group | Premenopausal Women: Progesterone Then Placebo | Premenopausal Women: Placebo Then Progesterone | Postmenopausal Women: Progesterone Then Placebo | Postmenopausal Women: Placebo Then Progesterone
Started | 9 | 9 | 3 | 6
Completed | 7 | 9 | 2 | 5
Not Completed | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — COVID-19 pandemic | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Premenopausal women: 18 participants were enrolled. Two participants were excluded from the outcome measures analysis because they did not complete all treatment phases (n=2). Thus 16 participants composed the final sample size for analysis of outcome measures. For analysis of adverse events, 18 participants received progesterone, and 16 participants received placebo; 16 participants received Ibutilide during the progesterone phase and 16 participants received ibutilide during placebo phase.
Groups:
- Premenopausal Women - Progesterone Then Placebo: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days. After a median 41-day washout period, participants received oral placebo, two capsules once daily every evening for 7 days.
- Premenopausal Women - Placebo Then Progesterone: Participants received oral placebo, two capsules once daily every evening for 7 days. After a median 41-day washout period, participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days.
- Postmenopausal Women - Progesterone Then Placebo: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days. After a washout period of at least two weeks, participants received oral placebo, two capsules once daily every evening for 7 days.
- Postmenopausal Women - Placebo Then Progesterone: Participants received oral placebo, two capsules once daily every evening for 7 days. After a washout period of at least two weeks, participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days.
- Total: Total of all reporting groups
Arm/Group | Premenopausal Women - Progesterone Then Placebo | Premenopausal Women - Placebo Then Progesterone | Postmenopausal Women - Progesterone Then Placebo | Postmenopausal Women - Placebo Then Progesterone | Total
Number analyzed (Participants) | 9 | 9 | 3 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6) | 29 (6) | 65 (4) | 64 (9) | 47 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 3 | 6 | 27
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 5 | 1 | 4 | 15
  Black | 2 | 2 | 2 | 2 | 8
  Asian | 2 | 2 | 0 | 0 | 4
  Hispanic | 1 | 1 | 0 | 0 | 2
  Non-Hispanic | 8 | 8 | 3 | 6 | 25
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 3 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Baseline (Pre-ibutilide) QT-F Intervals
Description: QT intervals will be corrected for heart rate using the Fridericia method
Time Frame: After 7 days of treatment with oral progesterone or placebo, prior to receiving ibutilide
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Premenopausal Women: Progesterone; Postmenopausal Women: Progesterone: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Progesterone: Participants received oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
- Premenopausal Women: Placebo; Postmenopausal Women: Placebo: Participants received oral placebo, two capsules once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms | 417 (11) | 421 (10) | 413 (21) | 414 (22)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.07, Mixed Models Analysis

2. Primary Outcome: Maximum Post-ibutilide QT-F Intervals
Description: Maximum post-ibutilide QT-F intervals
Time Frame: Prior to ibutilide; at 5 minutes into the 10-minute ibutilide infusion; end of infusion; and at 5, 10, 15, 20, 30, and 45 minutes and 1, 2, 4, 6, and 8 hours after the ibutilide infusion
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms | 465 (13) | 475 (9) | 450 (27) | 460 (28)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis

3. Primary Outcome: % Change From Baseline (Pre-ibutilide) in Maximum QT-F Intervals
Description: % change from baseline (pre-ibutilide) in maximum QT-F intervals
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline value
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
% change from baseline value | 11.3 (2.2) | 12.4 (2.5) | 9.2 (1.3) | 11.0 (3.0)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.16, Mixed Models Analysis

4. Primary Outcome: Area Under the QT-F Versus Time Curves During and for 1 Hour Following Ibutilide Infusion
Description: Area under the QT-F versus time curves during and for 1 hour
Time Frame: Prior to ibutilide; at 5 minutes into the 10-minute ibutilide infusion; end of infusion; and at 5, 10, 15, 20, 30, and 45 minutes and 1 hour after the ibutilide infusion
Measure: Mean (Standard Deviation); unit: ms*hr
Groups:
- Premenopausal Women: Progesterone; Postmenopausal Women: Progesterone: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Progesterone: Participants receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms*hr | 500 (13) | 510 (9) | 480 (33) | 510 (28)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis

5. Secondary Outcome: Baseline (Pre-ibutilide) Heart Rate-corrected J-Tpeak (J-Tpeakc) Intervals
Description: Baseline (pre-ibutilide) heart rate-corrected J-Tpeak (J-Tpeakc) intervals
Time Frame: After 7 days of treatment with oral progesterone or placebo, prior to receiving ibutilide
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms | 218 (25) | 221 (26) | 219 (10) | 219 (11)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.20, Mixed Models Analysis

6. Secondary Outcome: Maximum Post-ibutilide J-Tpeakc Intervals
Description: Maximum post-ibutilide J-Tpeakc intervals
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms | 230 (31) | 272 (28) | 234 (15) | 243 (13)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.01, Mixed Models Analysis

7. Secondary Outcome: % Change From Baseline (Pre-ibutilide) in Maximum J-Tpeakc Intervals
Description: % change from baseline (pre-ibutilide) in maximum J-Tpeakc intervals
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline value
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
% change from baseline value | 11.7 (5.8) | 14.1 (5.8) | 6.1 (3.5) | 7.9 (1.3)

8. Secondary Outcome: Area Under the J-Tpeakc Versus Time Curve During and for 1 Hour Following Ibutilide Infusion
Description: Area under the J-Tpeakc versus time curve during and for 1 hour following
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: ms*hr
Groups:
- Postmenopausal Women - Progesterone Then Placebo: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Progesterone: Participants received oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
- Postmenopausal Women - Placebo Then Progesterone: Participants received oral placebo, two capsules once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women - Progesterone Then Placebo | Postmenopausal Women - Placebo Then Progesterone
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms*hr | 248 (42) | 276 (40) | 258 (13) | 261 (14)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.015, Mixed Models Analysis

9. Secondary Outcome: Baseline (Pre-ibutilide) Tpeak-Tend Intervals
Description: Baseline (pre-ibutilide) Tpeak-Tend intervals
Time Frame: After 7 days of treatment with oral progesterone or placebo, prior to receiving ibutilide
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Postmenopausal Women - Placebo: Participants received oral placebo, two capsules once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women - Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms | 85 (6) | 88 (5) | 79 (8) | 80 (8)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.0005, Mixed Models Analysis

10. Secondary Outcome: Maximum Post-ibutilide Tpeak-Tend Intervals
Description: Maximum post-ibutilide Tpeak-Tend intervals
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Postmenopausal Women - Progesterone: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Progesterone: Participants received oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women - Progesterone | Postmenopausal Women - Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms | 99 (6) | 102 (5) | 81 (8) | 87 (9)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.017, Mixed Models Analysis

11. Secondary Outcome: % Change From Baseline (Pre-ibutilide) Maximum Tpeak-Tend Intervals
Description: % change from baseline (pre-ibutilide) maximum Tpeak-Tend intervals
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline value
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women - Progesterone | Postmenopausal Women - Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
% change from baseline value | 16.1 (5.6) | 16.0 (5.2) | 8.8 (3.6) | 10.5 (3.3)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p = 0.83, Mixed Models Analysis

12. Secondary Outcome: Area Under the Tpeak-Tend Versus Time Curves During and for 1 Hour Following Ibutilide Infusion
Description: Area under the Tpeak-Tend versus time curves during and for 1 hour following ibutilide infusion
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: ms*hr
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women - Progesterone | Postmenopausal Women - Placebo
Number analyzed (Participants) | 16 | 16 | 7 | 7
ms*hr | 98 (6) | 104 (7) | 90 (9) | 97 (9)
Statistical Analysis 1: Comparison: Premenopausal Women: Progesterone vs Premenopausal Women: Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Premenopausal women: During 7 days of therapy with progesterone and placebo, administered in randomized order, separated by a washout period. n=18 women completed the progesterone phase, n=16 women completed the placebo phase. Postmenopausal women: During 7 days of therapy with progesterone and placebo, administered in randomized order, separated by a washout period. n=7 women completed the progesterone phase, n=7 women completed the placebo phase.
Groups:
- Postmenopausal Women: Placebo: Participants received treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Progesterone: Participants received oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all participants to moderately lengthen the QT interval
Arm/Group | Premenopausal Women: Progesterone | Premenopausal Women: Placebo | Postmenopausal Women: Progesterone | Postmenopausal Women: Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 11/18 | 2/16 | 4/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premenopausal Women: Progesterone (N=18) | Premenopausal Women: Placebo (N=16) | Postmenopausal Women: Progesterone (N=7) | Postmenopausal Women: Placebo (N=7)
Fatigue/malaise (General disorders) | 7 (7) | 2 (2) | 4 (4) | 0 (0)
Spotting (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT03834883/Prot_SAP_000.pdf